CLINICAL TRIAL: NCT04076657
Title: Brock String Therapy for Receded Near Point of Convergence Post Concussion
Brief Title: Efficacy of Brock String Therapy Post Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Alicia Trbovich, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19070375
Record Dates: First submitted 2019-08-27; First posted 2019-09-03 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Concussion, Brain; Near Point Convergence
Keywords: brock string; sport-concussion; concussion therapy; receded near point of convergence
MeSH Terms: conditions — Brain Concussion | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care provider will not be aware of group assignment; participant will be aware of receiving treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brock String (Experimental): Participants will receive instruction on Brock String therapy after first clinic visit (<48 hours post) injury, and will complete home therapy exercise twice daily
  Interventions: Behavioral: Brock String Therapy
- Standard of Care (Active Comparator): Participants will receive standard of care (i.e., no Brock String therapy within the first week post injury) but will be informed they will receive any therapy deemed necessary at follow up visit 7-10 days post injury, consistent with standard of care
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Brock String Therapy — Oculomotor exercise to improve binocular vision function
  Arms: Brock String
Behavioral: Standard of Care — patient engages in normal behavior to manage vision issues, such as breaks with reading and screen use
  Arms: Standard of Care

SUMMARY:
The purpose of the proposed study is to evaluate the efficacy of Brock String therapy prescribed in the acute stage of concussion recovery can improve clinical outcomes among patients with receded near point of convergence (NPC).

Aim 1: Determine if participants receiving the Brock String have more significant improvements in NPC measurements at follow up 7-10 days post injury.

Aim 2: Determine if participants receiving the Brock String 1) improve on computerized neurocognitive test scores from initial visit (<48 hours post injury) to follow up visit (7-10 days post injury) compared to control participants, and 2) have reduced recovery time (i.e., days from injury until return to play) compared to control participants.

DETAILED DESCRIPTION:
Receded near point of convergence (NPC) is a common oculomotor deficit associated with numerous vision diagnoses, including convergence and accommodative insufficiencies, following sport-related concussion (SRC). Researchers have found associations with worse neurocognitive test scores, higher post-concussion symptom burden, and longer recovery among patients with receded NPC relative to concussion patients with normal NPC. Although oculomotor dysfunction may resolve spontaneously or improves with vision therapy exercises in the post-acute phase of recovery, it is unclear if early intervention can improve recovery outcomes. The Brock String is a cost effective and practical vision therapy exercise for congenital convergence insufficiency (CI), and initial research supports effectiveness with SRC patients who have receded NPC in the subacute phase of recovery (e.g., weeks to months post injury). Early vision therapy intervention may be efficacious in improving recovery times and reduce healthcare costs by eliminating later therapies for chronic deficits.

ELIGIBILITY:
Inclusion Criteria:

* Athletes who sustained a concussion during organized sport within past 48 hours
* ages 12-20
* at least one NPC measurement >10 centimeters at initial clinic evaluation.

Exclusion Criteria:

* lack of access to a smart phone to receive text message prompts
* vestibular disorder
* seizure disorder
* history of traumatic brain injury with imaging findings or brain surgery
* history of 3+ concussions\
* concussion within the past 6 months
* history of developmental or intellectual disability
* history of substance abuse
* Patients will also be excluded from recruitment if the treating clinician feels the potential participant would be unable to tolerate Brock String therapy due to severe symptoms

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Near point of convergence measurement | from visit 1 (<48 hours post injury) to visit 2 (7-10 days post injury)
  change in convergence measurement from nose in centimeters

SECONDARY OUTCOMES:
Immediate Post Concussion Assessment and Cognitive Testing (ImPACT | from visit 1 (<48 hours post injury) to visit 2 (7-10 days post injury)
  change in test scores based on normative data percentile (range <1-100); for all composite scores, including verbal memory, visual memory, visual motor speed scores, reaction time; better score indicating better performance
concussion recovery duration | from day of injury until final clinic visit, determined by concussion symptoms resolving and all aspects of testing within normal limits; expected range 7-10 days to up to 6 months post injury
  recovery time (i.e., days from injury until return to play)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Trbovich, PhD, Principal Investigator — University of Pittsburgh; Anthony P Kontos, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Rooney Sports Complex, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trbovich AM, Zynda AJ, Togashi T, Burley C, Mucha A, Collins MW, Kontos AP. Randomized Controlled Trial of Brock String Vision Therapy for Receded Near Point of Convergence Following Concussion. J Neurotrauma. 2025 Oct;42(19-20):1708-1718. doi: 10.1177/08977151251359960. Epub 2025 Sep 16. PMID 40957852